CLINICAL TRIAL: NCT00021229
Title: A Phase I/II Trial Of STI571 In Children With Newly Diagnosed Poor Prognosis Brainstem Gliomas And Recurrent Intracranial Malignant Gliomas
Brief Title: Imatinib Mesylate With or Without Radiation Therapy in Treating Young Patients With Newly Diagnosed or Recurrent Glioma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03019; PBTC-006 (Other: Pediatric Brain Tumor Consortium Protocol Identifier); U01CA081457 (NIH); CDR0000068761 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Results first posted 2010-04-09 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood central nervous system germ cell tumor; childhood high-grade cerebral astrocytoma; untreated childhood brain stem glioma; recurrent childhood brain stem glioma; recurrent childhood cerebral astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imatinib mesylate (Experimental)
  Interventions: Drug: imatinib mesylate; Radiation: local irradiation therapy

INTERVENTIONS:
Drug: imatinib mesylate — * Phase 1 Stratum I: Starting dose level of 350 mg/m2/day every 28 days X 13 courses (dose escalation)
  * Phase I Stratum IIA: Starting dose level of 465 mg/m2/day every 28 days X 13 courses (dose escalation)
  * Phase I Stratum IIB: Starting dose level of 465 mg/m2/day every 28 days X 13 courses (dose escalation)
  * Phase II: Phase I Stratum I determined dose (Maximum tolerated dose) every 28 days X 13 courses.
Radiation: local irradiation therapy — * Phase I Stratum I: Total dose of 5580 cGy using conventional or conformal volume-based delivery techniques once daily, 5 days/week for six weeks prior to receiving imatinib.
  * Phase II: Total dose of 5580 cGy using conventional or conformal volume-based delivery techniques once daily, 5 days/week for six weeks prior to receiving imatinib.

SUMMARY:
Phase I/II trial to estimate the maximum tolerated dose of imatinib mesylate in newly diagnosed brain stem gliomas and recurrent high grade gliomas and to assess the effectiveness of imatinib mesylate in treating young patients who have newly diagnosed intrinsic brain stem glioma. Imatinib mesylate may interfere with the growth of tumor cells by blocking the enzymes necessary for their growth. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining imatinib mesylate with radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of imatinib mesylate after completion of radiation in children with newly diagnosed poor prognosis brainstem gliomas. (Phase I, strata I closed to accrual as of 5/28/04.) II. Determine the maximum tolerated dose (MTD) of imatinib mesylate in children with recurrent high-grade intracranial glioma stratified according to the use of enzyme-inducing anticonvulsant drugs (EIACDs). (Phase I, strata IIA and IIB closed to accrual as of 8/15/03 and 8/15/04, respectively) III. Determine the safety and efficacy of this drug in patients with newly diagnosed diffuse intrinsic brainstem gliomas. (Phase II)

SECONDARY OBJECTIVES:

I. Explore neuroimaging and biological correlatives of therapeutic activity of this regimen in these patients. (Phase I, all strata closed to accrual as of 8/15/04) II. Determine the pharmacokinetics of these regimens in these patients overall and by enzyme-inducing anticonvulsant drugs (EIACDs) (Phase I, all strata closed to accrual as of 8/15/04.) III. Estimate the progression-free survival (PFS) and overall survival (OS) of newly diagnosed diffuse intrinsic brainstem gliomas treated with this drug. (Phase I and II)

OUTLINE: This is a phase I dose-escalation, multicenter study followed by a phase II. Patients are stratified according to tumor type (newly diagnosed intrinsic brainstem glioma vs recurrent/refractory intracranial high-grade glioma). Patients in stratum II (phase I only) are further stratified according to concurrent use of enzyme-inducing anticonvulsant drugs (EIACDs) (yes vs no). Patients are assigned to one of three strata in the phase I study.

* Phase I

  * Stratum I (newly diagnosed brainstem glioma): Patients undergo radiotherapy once daily five days a week for 6 weeks. Beginning 1-3 weeks after completion of radiotherapy, patients without evidence of intratumoral bleed receive oral imatinib mesylate twice daily. Imatinib mesylate treatment repeats every 4 weeks for up to 13 courses in the absence of disease progression or unacceptable toxicity. (Closed to accrual as of 5/28/04.)
  * Stratum II A (recurrent or refractory high-grade intracranial gliomas/no concurrent EIACDs): Patients receive imatinib mesylate as in stratum I. (Closed to accrual as of 8/15/03.)
  * Stratum II B (recurrent or refractory high-grade intracranial gliomas and concurrent EIACDs): Patients receive imatinib mesylate as in stratum I. (Closed to accrual as of 8/15/04.)

Cohorts of 2-3 patients receive escalating doses of imatinib mesylate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which it is estimated that 20% of patients will experience dose-limiting toxicity. MTDs are independently estimated in each strata. For stratum I, newly diagnosed brain stem gliomas, the dose level which at least 5 of 6 patients experience no dose-limiting toxicity will be the dose used in the efficacy and safety phase (phase II).

* Phase II: (Open to accrual as of 5/28/04.)

  * Stratum I only: Patients undergo radiotherapy as in phase I. Patients receive imatinib mesylate at the MTD established in phase I.

Patients enrolled in the phase I portion and not treated at the MTD are to be followed for the shortest of 1) three months after the last protocol based treatment or 2) the date other therapy is initiated. Stratum I patients treated at the MTD in the phase I portion and all patients in the phase II portion of the study are to be followed until death or withdrawal from the study

PROJECTED ACCRUAL: Approximately 140 patients will be accrued for this study within 2 years.

ELIGIBILITY:
Inclusion Criteria

* Age 3 to 21
* Performance status of Karnofsky 50-100% OR Lansky 50-100%
* Absolute neutrophil count greater than 1,000/mm3
* Platelet count greater than 100,000/mm3 (transfusion independent)
* Hemoglobin greater than 8 g/dL (transfusion allowed)
* Bilirubin no greater than 1.5 times normal for age
* SGPT less than 3 times normal for age
* Albumin at least 2 g/dL
* Creatinine less than 1.5 times normal for age OR Glomerular filtration rate greater than 70 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 6 months after study participation
* Stratum I

  * Newly diagnosed diffuse intrinsic brainstem malignant glioma
  * No disseminated disease
  * No radiographic evidence of intratumoral hemorrhage before or during radiotherapy
  * No prior chemotherapy (beyond routine corticosteroids)
  * No prior irradiation
  * Must not be receiving enzyme-inducing anticonvulsant drugs
* Stratum II

  * Histologically confirmed recurrent or refractory anaplastic astrocytoma, glioblastoma multiforme, or other high-grade glioma (including recurrent brain stem glioma
  * No intratumoral hemorrhage unrelated to prior surgical procedure
  * No myelosuppressive chemotherapy within 3 weeks (6 weeks if a nitrosourea agent) of study entry
  * No prior imatinib mesylate
  * At least 3 months since prior craniospinal radiotherapy (18 Gy or more)
  * At least 8 weeks since prior local radiotherapy to primary tumor
  * At least 2 weeks since prior focal radiotherapy for symptomatic
  * At least 3 months since prior bone marrow transplantation
  * Neurological deficits allowed if stable for at least 1 week prior to study

Exclusion Criteria

* Receiving other anticancer or experimental drug therapy.
* Ongoing uncontrolled infection.
* Significant cardiac, hepatic, gastrointestinal, renal, pulmonary, or psychiatric disease.
* Deep venous or arterial thrombosis within 6 weeks of registration.
* Taking warfarin.
* Newly diagnosed diffuse intrinsic brainstem malignant glioma with disseminated disease (stratum I)
* Intratumoral hemorrhage

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2001-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian F. Pollack, MD, Study Chair — University of Pittsburgh
Locations (10):
- United States (10):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Cancer Center and Hematology Service at Texas Children's Hospital, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington

REFERENCES:
- [Result] Williams G, Fahey FH, Treves ST, Kocak M, Pollack IF, Boyett JM, Kun LE, Poussaint TY. Exploratory evaluation of two-dimensional and three-dimensional methods of FDG PET quantification in pediatric anaplastic astrocytoma: a report from the Pediatric Brain Tumor Consortium (PBTC). Eur J Nucl Med Mol Imaging. 2008 Sep;35(9):1651-8. doi: 10.1007/s00259-008-0780-7. Epub 2008 Apr 19. PMID 18425516
- [Result] Pollack IF, Jakacki RI, Blaney SM, Hancock ML, Kieran MW, Phillips P, Kun LE, Friedman H, Packer R, Banerjee A, Geyer JR, Goldman S, Poussaint TY, Krasin MJ, Wang Y, Hayes M, Murgo A, Weiner S, Boyett JM. Phase I trial of imatinib in children with newly diagnosed brainstem and recurrent malignant gliomas: a Pediatric Brain Tumor Consortium report. Neuro Oncol. 2007 Apr;9(2):145-60. doi: 10.1215/15228517-2006-031. Epub 2007 Feb 9. PMID 17293590

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from PBTC member institutions were enrolled on the phase I component between 09May2001 and 28MAY2004 (stratum I), 15AUG2003 (stratum IIA), and 15AUG2004 (stratum IIB). The phase II component of the study opened on 28MAY2004 and was terminated on 13APR2005 due to poor accrual.
Pre-assignment Details: The intent of the phase I part of the study was to estimate the maximum tolerated dose (MTD) independently in stratum I, in stratum IIA, and in stratum IIB. The estimated MTD from stratum I was the recommended dose for the phase II part. Phase I participants in stratum I who received study drug at the MTD contributed to the phase II objectives.
Groups:
- Stratum I: Radiation + Imatinib Mesylate: Children with newly diagnosed brainstem gliomas received imatinib twice daily at a starting dose of 200 mg/m2/day. Treatment cycles were 4 weeks (maximum tolerated dose (MTD) estimation period - first 8 weeks) and imatinib was continued for up to 52 weeks in the absence of progression or serious toxicity.
  Local irradiation (RT) was administered concurrently with imatinib at the initiation of treatment with conventional fractionation at 180 cGy/day fractions, five days per week for six weeks, to a total dose of 5580 cGy.
  Because of concerns of intratumoral hemorrhage during RT, the protocol was amended (08JAN2003) to enroll patients without evidence of hemorrhage prior to RT and begin imatinib treatment 2 weeks (± 1 week) after completion of RT.
  Participants enrolled to the phase II part received imatinib at the MTD (from phase I) after RT.
  Six participants were enrolled on the phase I before the amendment, 29 after the amendment, and 1 on the phase II.
- Stratum IIA: Imatinib Mesylate: Children with recurrent high-grade gliomas not on enzyme-inducing anticonvulsant drugs (EIACDs) received imatinib twice daily at a starting dose of 350 mg/m2/day. Treatment cycles were 4 weeks (maximum tolerated dose (MTD) estimation period - first 4 weeks) and imatinib was continued for up to 52 weeks in the absence of progression or serious toxicity. Study participants did not receive radiation therapy in this stratum.
  Because of concerns of intratumoral hemorrhage, the protocol was amended (08JAN2003) to extend the MTD estimation period to 8 weeks (courses 1 and 2).
  Ten participants were enrolled on the phase I before the amendment and 23 after the amendment.
- Stratum IIB: Imatinib Mesylate: Children with recurrent high-grade gliomas on enzyme-inducing anticonvulsant drugs (EIACDs) received imatinib twice daily at a starting dose of 350 mg/m2/day. Treatment cycles were 4 weeks (maximum tolerated dose (MTD) estimation period - first 4 weeks) and imatinib was continued for up to 52 weeks in the absence of progression or serious toxicity. Study participants did not receive radiation therapy in this stratum.
  Because of concerns of intratumoral hemorrhage, the protocol was amended (08JAN2003) to extend the MTD estimation period to 8 weeks (courses 1 and 2).
  Eight participants were enrolled on the phase I before the amendment and eight after the amendment.
Period: Overall Study
Arm/Group | Stratum I: Radiation + Imatinib Mesylate | Stratum IIA: Imatinib Mesylate | Stratum IIB: Imatinib Mesylate
Started | 36 | 33 | 16
Enrolled in Phase I | 35 | 33 | 16
Maximum Tolerated Dose (MTD) Estimation | 23 (12 participants enrolled in the Phase I part did not complete the 8 week MTD estimation period.) | 20 (13 participants enrolled in the Phase I part did not complete the 8 week MTD estimation period.) | 12 (4 participants enrolled in the Phase I part did not complete the 8 week MTD estimation period.)
Enrolled in Phase II | 14 (Thirteen participants treated at the MTD in the phase I were also part of the phase II.) | 0 (Participants from stratum IIA did not participate in the phase II part of the study.) | 0 (Participants from stratum IIB did not participate in the phase II part of the study.)
Completed | 1 (1 participant completed 13 courses of therapy) | 0 | 0
Not Completed | 35 | 33 | 16
Not completed — Adverse Event | 10 | 5 | 2
Not completed — Death | 0 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 7 | 1
Not completed — Progressive Disease | 15 | 19 | 12
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Punctate hemmorrhage post RT | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum I: Radiation + Imatinib Mesylate | Stratum IIA: Imatinib Mesylate | Stratum IIB: Imatinib Mesylate | Total
Number analyzed (Participants) | 36 | 33 | 16 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36 | 30 | 15 | 81
  Between 18 and 65 years | 0 | 3 | 1 | 4
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.05 (4.3) | 10.9 (5.4) | 14.1 (4.7) | 10.3 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 9 | 47
  Male | 18 | 13 | 7 | 38
Region of Enrollment [Number; unit: participants]
  United States | 36 | 33 | 16 | 85

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Phase I Stratum I With Dose Limiting Toxicities (DLT) Observed During First 8 Weeks (Courses 1 and 2) of Imatinib Therapy
Description: The dose limiting toxicity (DLT) analysis population consists of phase I stratum I participants who developed DLT during the maximum tolerated dose (MTD) estimation period (course 1 and 2) or who completed the MTD estimation period (courses 1 and 2) without DLTs. DLTs observed during courses 1 and 2 were used to estimate the MTD. The estimated MTD based on the 23 participants who either had a DLT during course 1 or 2 or completed courses 1 and 2 without DLT is 265 mg/m2/day.
Time Frame: Day 1 of Imatinib Mesylate Therapy to Week 8
Population: Per protocol, participants included phase I stratum I participants who developed dose-limiting toxicities during the maximum tolerated dose (MTD) estimation period (courses 1 and 2) or who completed the MTD estimation period (courses 1 and 2) without dose-limiting toxicities.
Measure: Number; unit: Participants
Arm/Group | Stratum I: Radiation + Imatinib Mesylate
Number analyzed (Participants) | 23
Participants | 5

2. Primary Outcome: Number of Participants in Phase I Stratum II With Dose Limiting Toxicities (DLT) Observed During First 8 Weeks (Courses 1 and 2) of Imatinib Therapy
Description: The dose limiting toxicity (DLT) analysis population consisted of phase I stratum II participants who developed DLT during the maximum tolerated dose (MTD) estimation period (courses 1 and 2) or who completed the MTD estimation period (courses 1 and 2) without DLTs. DLTs observed during courses 1 and 2 were used to estimate the MTD. The estimated MTD based on the DLT analysis population of 20 in stratum IIA was 465 mg/m2/day. An MTD was not established in stratum IIB as no DLTs were observed at the higher dose levels of 620 and 800 mg/m2/day.
Time Frame: Day 1 of Imatinib Mesylate Therapy to Week 8
Population: Per protocol, participants included phase I stratum II participants who developed dose-limiting toxicities (DLT) during the maximum tolerated dose (MTD) estimation period (courses 1 and 2) or who completed the MTD estimation period (courses 1 and 2) without DLTs.
Measure: Number; unit: Participants
Arm/Group | Stratum IIA: Imatinib Mesylate | Stratum IIB: Imatinib Mesylate
Number analyzed (Participants) | 20 | 12
Participants | 2 | 0

3. Primary Outcome: Median Progression-free Survival (PFS)
Description: Progression-free survival is defined as the interval from initiation of treatment to the earliest of disease progression (tumor increase of 25% over baseline tumor measurement; appearance of new lesion(s); or progressive/worsening neurological status) or death for patients who failed, or to the last date of follow up for patients without failure.
Time Frame: Assessed pre-radiation, before the first dose of imatinib, and then every 8 weeks
Population: Per protocol, 40 participants who received at least one dose of drug were needed for this objective. The analysis population consists of stratum I participants enrolled at the maximum tolerated dose (phase 1) and the participants enrolled to the phase II part. The study was terminated because of poor accrual and the objective was not met.
Arm/Group | Stratum I: Radiation + Imatinib Mesylate
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline in Volume FLAIR at Two Weeks After Completion of Radiation
Description: This study attempted to investigate in an exploratory manner the effect of radiation (RT) on changes in various neuroimaging variables in pediatric brainstem gliomas (stratum I). Neuroimaging changes may have some association with outcome (response, survival, etc.). Volume FLAIR is one parameter obtained from standard magnetic resonance imaging (MRI) studies of the brain. Volume FLAIR was obtained at baseline (pre-radiation) and within two (+/- one) weeks after completion of RT.
Time Frame: Baseline and two weeks post completion of radiation
Population: The analysis population consists of Stratum I patients enrolled who had both pre and post radiation (RT) volume FLAIR measures. Stratum II participants did not receive RT and thus were not included.
Measure: Mean (Full Range); unit: cubic centimeters
Arm/Group | Stratum I: Radiation + Imatinib Mesylate
Number analyzed (Participants) | 24
cubic centimeters | 7.62 [-17.95 to 41.32]

5. Secondary Outcome: Peak Concentration (Cmax)
Description: Peak concentration (cmax) is a pharmacokinetic measure defined as the highest concentration of a drug measured after the drug is administered. The cmax of imatinib mesylate on day 1 of course 1 is reported. Two milliliter (0.5 ml for children under the age of 5) blood samples were collected immediately prior to imatinib mesylate administration on Day 1 of Course 1 and at the following timepoints following drug administration: 0.5, 1, 1.5, 2, 4, 10 and 12 hours after the morning dose.
Time Frame: Day 1 of Course 1
Population: The analysis population consists of participants who enrolled at the maximum tolerated dose (MTD) of the phase I component and who submitted day 1 course 1 samples for the PK studies. An MTD was not estimated in stratum IIB. For this stratum, reported are values at the stratum IIA MTD to allow comparison.
Measure: Mean (Full Range); unit: µg/ml
Arm/Group | Stratum I: Radiation + Imatinib Mesylate | Stratum IIA: Imatinib Mesylate | Stratum IIB: Imatinib Mesylate
Number analyzed (Participants) | 3 | 9 | 3
µg/ml | 1.3 [.7 to 2.1] | 2.6 [1.5 to 5.9] | 1.3 [.8 to 2.1]

6. Secondary Outcome: Median Overall Survival
Description: Overall Survival (OS) is defined as the interval from initiation of treatment to death or date of last contact for surviving patients.
Time Frame: Assessed before radiation therapy, before the first dose of imatinib, then every 8 weeks.
Population: The analysis population consists of the stratum I participants who received imatinib mesylate at or above the maximum tolerated dose. The median survival reported is based on these 20 participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Stratum I: Radiation + Imatinib Mesylate
Number analyzed (Participants) | 20
Days | 324.5 (8.7) [216 to 383]

7. Secondary Outcome: Pre-treatment Basic Fibroblast Growth Factor Values From Urine
Description: This study attempted to investigate in an exploratory manner the effect of biological markers on tumor growth. Basic fibroblast growth factor (bFGF) may play a role in tumor development by helping tumor vessels establish and grow. Urine was collected from participants before treatment to measure the baseline urine bFGF values.
Time Frame: Pre-treatment
Population: Per protocol, the analysis population consists of participants treated on the phase I component who submitted pre-treatment urine samples for the biomarker study.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Stratum I: Radiation + Imatinib Mesylate | Stratum IIA: Imatinib Mesylate | Stratum IIB: Imatinib Mesylate
Number analyzed (Participants) | 16 | 17 | 10
pg/ml | 5665 (4006) | 10322 (14443) | 5312 (6262)

8. Secondary Outcome: Pre-treatment Basic Fibroblast Growth Factor Values From Plasma
Description: This study attempted to investigate in an exploratory manner the effect of biological markers on tumor growth. Basic fibroblast growth factor (bFGF) may play a role in tumor development by helping tumor vessels establish and grow. Blood (plasma) was drawn from participants before treatment to measure the baseline plasma bFGF values.
Time Frame: Pre-treatment
Population: Per protocol, the analysis population consists of participants treated on the phase I component who submitted pre-treatment blood samples for the biomarker study.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Stratum I: Radiation + Imatinib Mesylate | Stratum IIA: Imatinib Mesylate | Stratum IIB: Imatinib Mesylate
Number analyzed (Participants) | 19 | 16 | 10
pg/ml | 8.69 (7.16) | 32.3 (64.5) | 11.3 (12.2)

9. Secondary Outcome: Pre-treatment Vascular Endothelial Growth Factor From Urine
Description: This study attempted to investigate in an exploratory manner the effect of biological markers on tumor growth. Vascular endothelial growth factor (VEGF) may play a role in tumor development by helping tumor vessels establish and grow. Urine was collected from participants before treatment to measure the baseline urine VEGF values.
Time Frame: Pre-treatment
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Stratum I: Radiation + Imatinib Mesylate | Stratum IIA: Imatinib Mesylate | Stratum IIB: Imatinib Mesylate
Number analyzed (Participants) | 16 | 17 | 10
pg/ml | 79 (69.9) | 86.1 (93.9) | 45.3 (38.0)

10. Secondary Outcome: Pre-treatment Vascular Endothelial Growth Factor Values From Plasma
Description: This study attempted to investigate in an exploratory manner the effect of biological markers on tumor growth. Vascular endothelial growth factor (VEGF) may play a role in tumor development by helping tumor vessels establish and grow. Blood (plasma) was drawn from participants before treatment to measure the baseline plasma VEGF values.
Time Frame: Pre-treatment
Population: as for outcome 8
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Stratum I: Radiation + Imatinib Mesylate | Stratum IIA: Imatinib Mesylate | Stratum IIB: Imatinib Mesylate
Number analyzed (Participants) | 19 | 16 | 10
pg/ml | 119.9 (168.5) | 155.2 (229.7) | 78.2 (59.4)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed weekly during the first four weeks (course 1), every 2 weeks during the next 2 courses (8 weeks total), every 4 weeks for all subsequent courses (up to 13 courses), and through 30 days following the end of treatment.
Description: Assessments were made routinely for all patients per the schedule of clinical and laboratory assessments outlined in the protocol.
Arm/Group | Stratum I: Radiation + Imatinib Mesylate | Stratum IIA: Imatinib Mesylate | Stratum IIB: Imatinib Mesylate
Serious Adverse Events (participants affected / at risk) | 13/36 | 13/33 | 5/16
Other Adverse Events (participants affected / at risk) | 33/36 | 31/33 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum I: Radiation + Imatinib Mesylate (N=36) | Stratum IIA: Imatinib Mesylate (N=33) | Stratum IIB: Imatinib Mesylate (N=16)
Abdominal pain or cramping (Gastrointestinal disorders) | 1 | 1 | 0
Bicarbonate (Metabolism and nutrition disorders) | 1 | 0 | 0
CNS hemorrhage/bleeding (Nervous system disorders) | 7 | 7 | 2
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Confusion (Nervous system disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Creatinine (Renal and urinary disorders) | 1 | 0 | 0
Dehydration (Gastrointestinal disorders) | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 1 | 1
Diarrhea without colostomy (Gastrointestinal disorders) | 1 | 1 | 0
Edema (Blood and lymphatic system disorders) | 1 | 1 | 0
Fatigue (General disorders) | 2 | 3 | 0
Fever (in the absence of neutropenia) (General disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 3 | 3
Hematemesis (Vascular disorders) | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 0
Hypoalbuminemia (Hepatobiliary disorders) | 2 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Incontinence (Renal and urinary disorders) | 1 | 0 | 0
Infection without neutropenia (Infections and infestations) | 3 | 0 | 0
Inpatient Hospital Days (General disorders) | 1 | 0 | 0
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Melena/GI bleeding (Gastrointestinal disorders) | 0 | 1 | 0
Memory loss (Nervous system disorders) | 0 | 0 | 1
Metabolic/Laboratory- Other (Metabolism and nutrition disorders) | 1 | 0 | 0
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Neurology - Other (Nervous system disorders) | 1 | 1 | 0
Neuropathy - Motor (Nervous system disorders) | 1 | 1 | 1
Neuropathy - cranial (Nervous system disorders) | 1 | 0 | 0
Neuropathy - sensory (Nervous system disorders) | 1 | 0 | 0
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 | 1 | 0
Pain - other (General disorders) | 1 | 0 | 0
Pigmentation changes (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Platelets (Blood and lymphatic system disorders) | 0 | 1 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Renal/Genitourinary - Other (Renal and urinary disorders) | 2 | 0 | 0
Seizures (Nervous system disorders) | 1 | 0 | 1
Speech impairment (Nervous system disorders) | 1 | 1 | 0
Thrombosis/embolism (Blood and lymphatic system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum I: Radiation + Imatinib Mesylate (N=36) | Stratum IIA: Imatinib Mesylate (N=33) | Stratum IIB: Imatinib Mesylate (N=16)
Abdominal pain or cramping (Gastrointestinal disorders) | 8 | 2 | 2
Alkaline phosphatase (Investigations) | 1 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 10 | 5 | 1
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Ataxia (incoordination) (Nervous system disorders) | 8 | 5 | 3
Bicarbonate (Metabolism and nutrition disorders) | 4 | 3 | 0
Bilirubin (Hepatobiliary disorders) | 3 | 1 | 0
CNS hemorrhage/bleeding (Nervous system disorders) | 3 | 0 | 0
Cognitive/disturbance/learning problems (Nervous system disorders) | 1 | 1 | 1
Conjunctivitis (Eye disorders) | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 14 | 3 | 1
Constitutional symptoms - Other (General disorders) | 2 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Creatinine (Investigations) | 3 | 1 | 0
Cushingnoid appearance (Endocrine disorders) | 8 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 1 | 2
Dermatology/skin -Other (Skin and subcutaneous tissue disorders) | 4 | 5 | 1
Diarrhea without colostomy (Gastrointestinal disorders) | 7 | 6 | 1
Dizziness/light-headedness (Nervous system disorders) | 4 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Dyspepsia/heartburn (Gastrointestinal disorders) | 6 | 3 | 0
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 2 | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 0
Earache (otalgia) (Ear and labyrinth disorders) | 5 | 0 | 1
Edema (Vascular disorders) | 1 | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
External auditory canal (Ear and labyrinth disorders) | 2 | 0 | 0
Fatigue (General disorders) | 13 | 11 | 4
Fever (in the absence of neutropenia) (General disorders) | 5 | 2 | 0
Flatulence (Gastrointestinal disorders) | 2 | 1 | 0
GGT (Investigations) | 1 | 0 | 3
Gastrointestinal-Other (Gastrointestinal disorders) | 1 | 2 | 0
Headache (Nervous system disorders) | 18 | 16 | 9
Hemoglobin (Blood and lymphatic system disorders) | 17 | 10 | 7
Hepatic-Other (Hepatobiliary disorders) | 1 | 0 | 2
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 11 | 9 | 5
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 1 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 6 | 3 | 2
Hypernatremia (Metabolism and nutrition disorders) | 3 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypoalbuminemia (Hepatobiliary disorders) | 5 | 4 | 6
Hypocalcemia (Metabolism and nutrition disorders) | 10 | 7 | 5
Hypoglycemia (Metabolism and nutrition disorders) | 5 | 1 | 2
Hypokalemia (Metabolism and nutrition disorders) | 9 | 7 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 10 | 3 | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 16 | 10 | 6
Incontinence (Renal and urinary disorders) | 2 | 2 | 0
Infection without neutropenia (Infections and infestations) | 10 | 5 | 1
Infection/Febrile Neutropenia-Other (Infections and infestations) | 0 | 1 | 1
Inner ear/hearing (Ear and labyrinth disorders) | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 5 | 1 | 0
Irritability (<3 years of age) (General disorders) | 3 | 1 | 0
Leukocytes (Blood and lymphatic system disorders) | 18 | 9 | 6
Lymphopenia (Blood and lymphatic system disorders) | 19 | 8 | 7
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 5 | 1 | 2
Mood alteration - anxiety, agitation (Psychiatric disorders) | 3 | 1 | 0
Mood alteration - depression (Psychiatric disorders) | 2 | 3 | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0
Musculoskeletal-Other (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Nausea (Gastrointestinal disorders) | 12 | 10 | 7
Neurology - other (Nervous system disorders) | 3 | 3 | 0
Neuropathic pain (General disorders) | 1 | 2 | 0
Neuropathy - cranial (Nervous system disorders) | 7 | 3 | 0
Neuropathy - motor (Nervous system disorders) | 9 | 9 | 6
Neuropathy - sensory (Nervous system disorders) | 3 | 3 | 1
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 15 | 8 | 4
Nystagmus (Nervous system disorders) | 2 | 2 | 2
Ocular/Visual - Other (Eye disorders) | 1 | 3 | 0
Pain - other (General disorders) | 6 | 4 | 5
Personality/behavioral (Psychiatric disorders) | 2 | 2 | 1
Platelets (Blood and lymphatic system disorders) | 8 | 6 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0 | 1
Pulmonary-Other (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7 | 8 | 5
Renal/Genitourinary-Other (Renal and urinary disorders) | 0 | 2 | 1
SGOT (AST) (Hepatobiliary disorders) | 14 | 8 | 4
SGPT (ALT) (Hepatobiliary disorders) | 15 | 9 | 4
Seizure(s) (Nervous system disorders) | 1 | 4 | 5
Speech impairment (Nervous system disorders) | 5 | 2 | 1
Stomatitis/pharyngitis (Gastrointestinal disorders) | 3 | 2 | 1
Transfusions: pRBCs (Blood and lymphatic system disorders) | 0 | 1 | 1
Tremor (Nervous system disorders) | 3 | 2 | 1
Urinary frequency/urgency (Renal and urinary disorders) | 1 | 1 | 2
Urinary retention (Renal and urinary disorders) | 3 | 1 | 0
Vision - blurred vision (Eye disorders) | 2 | 2 | 0
Vision - double vision (Eye disorders) | 9 | 2 | 2
Vomiting (Gastrointestinal disorders) | 23 | 13 | 8
Weight gain (Investigations) | 5 | 4 | 1
Weight loss (Investigations) | 2 | 0 | 1
Rash/Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
The phase II component of the trial was terminated because of poor accrual. Only one patient enrolled to the phase II component and did not receive the investigational drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less